CLINICAL TRIAL: NCT00441688
Title: Prospective Epidemiological Study of the Prevalence of HLAB*5701 in HIV-1 Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Other
Other Study IDs: 109477
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Human Immunodeficiency virus; HLAgenetics polymorphism
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GI265235 (Experimental)
  Interventions: Drug: GI265235

INTERVENTIONS:
Drug: GI265235

SUMMARY:
This study is a cross sectional observational study to evaluate the prevalence of HLA-B*5701 in the major French ethnotypes.

Any HIV-1 infected subject will be eligible for this study including antiretroviral therapy (ART) naÃ-ve and experienced subjects irrespective of abacavir use, as well as subjects previously tested for HLA-B*5701. Subjects will be approached during a standard clinic visit, and all subjects will be consented prior to any study specific procedure. Subjects will be asked to provide a tissue sample (cheek cells and blood sample) which will be used to assess HLA-B*5701 status by central and local methodologies.

ELIGIBILITY:
Inclusion criteria:

* HIV-1 infected patients, ART naive or experienced over the age of 18 years.
* Patients must be either affiliated to or beneficiary of a social security category.
* Patient is willing and able to understand and provide written informed consent prior to participation in this study.

Exclusion criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2007-03-15 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2007-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with HLA-B*5701 in the French HIV-1 infected population assessed using centralized screening assay results | Day 1
  Tissue sample (cheek cells and blood sample) were collected from the participants to assess HLA-B*5701 status using centralized screening assay in the centralized laboratory.The prevalence was calculated as the ratio of the number of participants with HLA-B*5701 positive divided by the total number of participants with available HLAB*5701 result multiplied by 100.

SECONDARY OUTCOMES:
Percentage of participants with HLA-B*5701 in the major French ethnotypes in the study population | Day 1
  Participants attended a single visit where an assessment of the participant's demographic background (age, sex , mode of HIV transmission, ethnicity, country of origin and parental country of origin) was conducted, and tissue samples (buccal cells and blood sample) were collected to determine the presence of HLA-B*5701 genotype by both central and local laboratories using centralized screening assay. The prevalence was calculated as the ratio of the number of participants with HLA-B*5701 positive divided by the total number of subjects with available HLAB*5701 result multiplied by 100. Data is presented for the prevalence of HLA-B*5701 in all the ethnotypes.
Number of participants with positive HLA-B*5701 screening results obtained with local laboratory | Day 1
  Tissue sample (cheek cells and blood sample) were collected from the participants to assess HLA-B*5701 status using centralized screening assay in the local laboratory. The prevalence was calculated as the ratio of the number of participants with HLA-B*5701 positive divided by the total number of subjects with available HLAB*5701 result. According to local laboratory, participants with positive results have been summarized here.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare